CLINICAL TRIAL: NCT01288508
Title: Investigation of Supra Fiber in the Treatment of Adults With Constipation-A Double-blind Randomized Controlled Trial
Brief Title: Investigation of Supra Fiber in the Treatment of Adults With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Supra Fiber
Record Dates: First submitted 2011-01-19; First posted 2011-02-02 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Supra Fiber (Active Comparator)
  Interventions: Dietary Supplement: Supra Fiber
- Psyllium (Active Comparator)
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Dietary Supplement: Supra Fiber — 2 tablespoons of fiber taken with 8oz water taken twice a day for 30 days
  Arms: Supra Fiber
Dietary Supplement: Psyllium — 1 tablespoon of fiber taken with 8 oz water twice a day for 30 days
  Arms: Psyllium

SUMMARY:
Background: Whether Supra-Fiber, a plum-derived fiber supplement is useful in the treatment of constipation is not known. Supra Fiber is the first fiber supplement that has a blend of whole food fruit as its main ingredient. It contains prunes, pomegranates, blueberries, and Acai berries. Unlike psyllium, which is mostly (90%) insoluble fiber, Supra Fiber is a balanced (50%) blend of insoluble and soluble fiber. This may provide the beneficial effects of fiber, and eliminate potential adverse symptoms of fiber such as bloating, distention, hard bulky stools and excess gas. In this study, we expect to not only evaluate the efficacy but also the palatability and tolerability of Supra Fiber in the treatment of chronic constipation.

Aims:

1. To investigate and compare the effects of Supra Fiber (5 grams BID) or psyllium (5 grams BID) on the number of complete spontaneous bowel movements per week, and bowel symptoms.
2. To examine the effects of fiber supplements on taste and quality of life in adults with functional chronic constipation in a randomized, double-blind, parallel group controlled trial.

Methods: We propose to enroll 90 subjects with functional constipation in a single blinded, randomized, cross-over study comparing 4 weeks of Supra Fiber with 4 weeks of treatment with Psyllium

Data analysis: The primary outcome measure will be the global relief of constipation symptoms as rated by the subject at the end of each phase of the study. Additionally, we will assess several secondary outcome measures that will include the number of Complete Spontaneous Bowel Movements (CSBM) per week, Quality of Life , psychological profile, patient rating of taste on a VAS scale, patient rating of bloating, distension, satiety and fullness and patient rating of constipation-related symptoms.

Expected results: We anticipate that treatment with Supra Fiber will improve symptoms of constipation compared to the baseline. This improvement will be comparable or superior to that achieved with psyllium treatment. Additionally, Supra Fiber will offer a natural, food based, convenient and more tasty alternative to over-the-counter laxatives and fiber supplements.

ELIGIBILITY:
Inclusion Criteria:

* Constipation as defined by Rome III criteria (3,4). Also, patients should have insufficient criteria for IBS, and only rarely experience loose stools without the use of laxatives.
* Adults between the ages of 18-75 years

Exclusion Criteria:

* Patients taking drugs that are known to be constipating will be excluded or asked to discontinue medications for at least 2 weeks and reassessed. Patients who remain constipated will be eligible for enrollment.
* Co-morbid illnesses such as severe cardiovascular disease, chronic renal failure
* Previous gastrointestinal surgery except cholecystectomy and appendectomy.
* Neurologic diseases such as multiple sclerosis, strokes, spinal cord injuries, and those who have problems with cognizance, i.e. a mini-mental score of <15 and/or are legally blind
* Hirschsprung' s disease, or active local anorectal problems such as anal fissures, bleeding hemorrhoids,
* Alternating constipation and diarrhea and those who fulfill the Rome-III criteria for irritable bowel syndrome.
* Subjects with a known allergy to psyllium or plums.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of Complete Spontaneous Bowel Movements (CSBM) per week | 9 Weeks
  1. Number of Complete Spontaneous Bowel Movements (CSBM) per week. This will be analyzed from the daily stool diaries (Appendix 1). The CSBM provides a more robust and better assessment of the overall change in bowel function that takes into account not only the stool frequency but also the completeness and satisfaction with bowel function. A CSBM is defined as a bowel movement that is produced without the use of additional laxatives, suppositories or enemas in the previous 24 hours, other than the study medication.

SECONDARY OUTCOMES:
Global Relief of Constipation | 9 Weeks
  1. Global relief of constipation.
  2. Other Parameters of bowel function including stool frequency, stool consistency (Bristol Stool Scale), Straining effort, Feeling of complete evacuation, bloating, and distension

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States